CLINICAL TRIAL: NCT01750892
Title: Transition From Pediatric to Adult Services: A Primary Care Based Model for Patients With Chronic Conditions
Brief Title: Primary Care Transition Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Peter_12-009117
Record Dates: First submitted 2012-12-13; First posted 2012-12-17 (Estimated); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Chronic Health Condition; Cognitive Disability

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group 1: Control (Active Comparator): Group 1 will be the control group. They will complete questionnaires but will otherwise receive usual care from their Primary Care Provider (PCP). At the end of the study period they will be given the Study Materials for participating.
  Interventions: Other: Study Materials
- Group 3: Group Intervention (Experimental): Group 3 (Group Intervention) will receive the Study Materials at the beginning of the study and will also be invited to attend two REACH for Independence group sessions.
  Interventions: Behavioral: REACH for Independence; Other: Study Materials
- Group 4: Full Intervention (Experimental): Group 4 (Full Intervention) will receive the Study Materials at the beginning of the study, will be invited to attend the REACH for Independence group sessions, and will be invited to a Transition Consult with an MD and social worker.
  Interventions: Behavioral: REACH for Independence; Behavioral: Transition Consult; Other: Study Materials
- Group 2: Basic Intervention (Experimental): Group 2 (Basic Intervention) will receive the Study Materials at the beginning of the study but will otherwise continue with their usual PCP care.
  Interventions: Other: Study Materials

INTERVENTIONS:
Behavioral: REACH for Independence — REACH for Independence is a transition and self-care skill-building peer support group led by a social worker. It is comprised of two 2.5-hour group sessions where participants participate in activities designed to teach self-care, self-advocacy and improve transition to adulthood skills.
  Arms: Group 3: Group Intervention; Group 4: Full Intervention
Behavioral: Transition Consult — The transition consult is a 1-on-1 visit with an MD and social worker. At the consults, participants will receive individualized information related to their unique medical and psychosocial needs and support related to issues relevant to their gaining healthcare independence and finding an adult doctor, such as accommodations, transportation, insurance and finances. After the consult, this group will have access to a transition coordinator who can help with any transition-related problems that may occur.
  Arms: Group 4: Full Intervention
Other: Study Materials — The Study Materials include a Care Binder, a Resource list, an Adult Doctor List and a Wallet Card. The Care Binder is an organizational tool to help patients with special healthcare needs manage and track important information related to their health and medical care. The Resource list has information about important community resources. The Adult Doctor List provides information about finding an adult primary care provider. The Wallet Card is a sheet for tracking important medical and personal information.

SUMMARY:
This study is looking at ways to help young people with chronic health conditions take better care of their health and find an adult doctor.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether providing targeted transition-related skills through interventions with varying degrees of intensity (from the low intensity Basic intervention group, to the mild intensity Group Intervention group, to the high intensity Full Intervention group) results in improved transition readiness and self-care skills and improved successful transition to adult-based services for young adults with chronic health conditions. Secondary objectives include determining if the transition interventions enhance transition-related satisfaction among participants, their caregivers and the involved pediatric and adult providers.

ELIGIBILITY:
Young Adult Inclusion Criteria:

* Males or females age 19 years of age or older
* Presence of at least 1 Chronic Condition and/or Cognitive Disability
* Last visit with pediatric primary care provider occurring on or after January 1, 2011
* Currently active in one of four identified pediatric practices (Cobbs Creek, Chestnut Hill, Market Street, West Chester)
* Current primary care provider approval for participation
* English speaking

Young Adult Exclusion Criteria:

* Male or female age < 19 years
* No presence of a chronic condition or cognitive disability
* Last visit with pediatric PCP occurring prior to January 1, 2011
* Not currently active in one of four identified pediatric practices (Cobbs Creek, Chestnut Hill, Market Street, West Chester)
* Current PCP disapproves participation
* Non-English speaking

Caregiver Inclusion Criteria:

* Has a child enrolled in the study
* Child has consented/assented to allow them to participate
* English speaking

Caregiver Exclusion Criteria:

* Child did not consent/assent to allow them to participate
* Non-English speaking

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Successful transition to an adult provider | 10 months
  The primary outcome is successful transition to an adult provider, as evidenced by at least 1 visit with an adult provider within 10 months of the baseline visit.

SECONDARY OUTCOMES:
Increased self-care and transition related skills | 6 months
  Self-care and transition related skills will be measured pre- and post- intervention with the Transition Readiness Assessment Questionnaire (TRAQ). The TRAQ is a validated 33-item self-administered tool that measures skills needed to progress towards independence in key areas of life like education and work as well as skills needed to successfully transition from pediatric to adult healthcare. The TRAQ will be completed over the phone or via an online survey with young adult participants and their caregivers at baseline and at the 6-month follow-up visit.

OTHER OUTCOMES:
Participant satisfaction with the intervention | 6 months
  Self-reported satisfaction with the intervention will be assessed at 6-months post-baseline via a phone interview or online survey.

CONTACTS AND LOCATIONS:
Overall Officials: Nadja Peter, MD, Principal Investigator — Children's Hospital of Philadelphia; Oana Tomescu, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States